CLINICAL TRIAL: NCT05913141
Title: Patient-derived Organoids, Patient-derived Organoids-tumor-infiltrating Lymphocyte Coculture System, and Patient-derived Organotypic Tissue Spheroids for Drug Screen
Brief Title: PDO/PDO-TIL/PDOTS for Drug Screen
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hu Bo, Doctor, Shanghai Zhongshan Hospital
Other Study IDs: B2022-063R
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Liver Cancer; Metastatic Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Drug Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Patients tumor sample and peritumor sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with PDO/PDO-TIL/PDOTS: Patients whose tumors were established into patient-derived organoids, patient-derived organoids-tumor-infiltrating lymphocyte coculture systems, or patient-derived organotypic tissue spheroids, and screened for drug-sensitive.
  Interventions: Other: Drug screen with PDO/PDO-TIL/PDOTS

INTERVENTIONS:
Other: Drug screen with PDO/PDO-TIL/PDOTS — Drug screen with patient-derived organoids, patient-derived organoids-tumor-infiltrating lymphocyte coculture system, or patient-derived organotypic tissue spheroids.

SUMMARY:
This clinical trial aims to use the patient-derived organoid (PDO), Patient-derived organoids-tumor-infiltrating lymphocyte coculture system (PDO-TIL) and patient-derived organotypic tissue spheroids (PDOTS) to simulate the tumor microenvironment in cancer patients. The culture system can be used for pre-clinical validation of drugs and screening of drugs to treat sensitive people and provide individualized treatment for patients with liver cancer. This model is used to explore the molecular mechanism of drug resistance and to find intervention strategies to further improve the response rate of drugs. This study is expected to provide an ideal platform for drug screening and drug resistance research in liver cancer patients, which can replace experimental animal models, and guide personalized medication for liver cancer patients, so as to improve the overall prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, male or female.
2. Liver cancer or metastatic liver cancer diagnosed clinically or pathologically, at least one measurable lesion.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
4. Patient has given written informed consent.
5. The function of important organs meets the requirements.
6. Non-surgical sterilization or women of childbearing age need to use a medically-accepted contraceptive (such as an intrauterine device, contraceptive or condom) during the study period and within 3 months after the end of the study treatment period.

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid Hyperfunction; patients with vitiligo; complete remission of asthma in childhood, can be included without any intervention after adulthood; asthma patients who require bronchodilators for medical intervention cannot be included).
2. The patient is using immunosuppressive agents or systemic hormonal therapy to achieve immunosuppressive purposes (agents amount > 10 mg/day of prednisone or other therapeutic hormones), and continue to use within 2 weeks before enrollment.
3. Have clinical symptoms or diseases that are not well controlled.
4. Significant clinically significant bleeding symptoms or a clear bleeding tendency within 3 months prior to randomization.
5. Arterial/venous thrombosis in the first 6 months of randomization.
6. According to the investigator, the patient has other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, and serious laboratory abnormalities.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver cancer or metastatic liver cancer
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 years
  Evaluated by researchers based on the RECIST 1.1 standard

SECONDARY OUTCOMES:
Progression free survival (PFS) | Evaluated by researchers based on the RECIST 1.1 standard
  1 years
Relapse-free survival (RFS) | 1 year
  From the date of enrollment to tumor recurrence or Death
Overall survival (OS) | 1 years
  The date of Death of any causes since the date of enrollment
To the relief time (TOR) | 1 years
  Evaluated by researchers based on the RECIST 1.1 standard
Duration of relief (DOR) | 1 years
  Evaluated by researchers based on the RECIST 1.1 standard
Disease control rate (DCR) | 1 years
  Evaluated by researchers based on the RECIST 1.1 standard
6-month survival rate | 6 months
  Evaluated by researchers based on the RECIST 1.1 standard
12-month survival rate | 12 months
  Evaluated by researchers based on the RECIST 1.1 standard

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No